CLINICAL TRIAL: NCT01349335
Title: A Phase 2 Randomized, Double-blinded, Multicenter and Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of Different Doses of Tolvaptan Tablet in Patients With Cirrhotic Ascites
Brief Title: Dose Exploring and Setting Study for Tolvaptan to Treat Hepatic Cirrhosis With Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-08-804-01
Record Dates: First submitted 2010-03-05; First posted 2011-05-06 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2011-05

CONDITIONS: Ascites; Hepatic Cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. tolvaptan (Experimental): 15 mg, P.O., Qd, for 7 days,
  Interventions: Drug: Tolvaptan
- 2 tolvaptan (Experimental): 30 mg, P.O., Qd, for 7 days,
  Interventions: Drug: Tolvaptan
- 3. Placebo (Experimental): 30mg,P.O.,Qd, for 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tolvaptan — tablet, 15 mg, Qd, for 7 days
  Other Names: SAMSCA
  Arms: 1. tolvaptan
Drug: Tolvaptan — tablet, 30 mg, Qd, 7 days
  Other Names: SAMSCA
  Arms: 2 tolvaptan
Drug: placebo — tablet, 30 mg, Qd, 7days.
  Other Names: blank tablet
  Arms: 3. Placebo

SUMMARY:
To observe the safety/efficacy of tolvaptan for treatment of patients with hepatic cirrhosis with ascites and exploring the dosage-effect relations of the drug.

DETAILED DESCRIPTION:
Tolvaptan is able to exert hydragogue diuretic effects (water diuresis) via inhibition of water reabsorption by renal collecting ducts without corresponding increase in electrolyte excretion. It has been confirmed that tolvaptan is able to increase urine volume without any adverse effects on renal functions.

ELIGIBILITY:
Inclusion Criteria:

1. hepatic cirrhosis patients after 7days treatment of loop diuretics and aldosterone antagonist but still with ascites
2. Hospitalized patients or those who can be hospitalized in this trial between observation period and posttherapeutic observation (Visits at clinic will be allowed after day 8);
3. During the observation period (-3 day to -1 day ), subjects whose body weight difference fall within ±1.0 kg range 2 days (day-2 and day -1) prior to initiation of trial drug treatment;
4. Ages: ≥18 and ≤75 years of age;
5. Genders: men or women;
6. Signed the Informed Consent Form.

Exclusion Criteria:

1. Patients with the following diseases, complications or symptoms:

   * Hepatic encephalopathy (Coma scale Note 1) grade 2 or higher);
   * Malignant ascites;
   * Uncontrolled spontaneous bacterial peritonitis;
   * Patients are likely to experience alimentary tract hemorrhage during the trial;
   * Heart failure (NYHA cardiac function scale Note 2) stages 3 and 4);
   * Anuria (daily urine volume below 100mL);
   * Dysuria resulting from urethral stricture, calculus and tumors.
2. Patients with the following medical history:

   * Alimentary tract hemorrhage within 10 days prior to screening;
   * Cerebrovascular accident within 1 month prior to screening;
   * Gout attack within 1 month prior to screening;
   * Past allergy or hypersensitive reactions to benzodiazepines (e.g. benazepril hydrochloride)
3. Systolic pressure below 90mmHg at screening;
4. Patients with the following abnormalities in laboratory examinations at screening:

   Serum creatinine exceeds 2.5X upper limits of normal, serum Na+>145mmol/L (or exceeds upper limits of normal), serum K+>5.5mmol/L, uric acid>8.0mg/dL (476μmol/L), Child-pugh scale greater than 12.
5. Patients cannot take drugs orally;
6. Pregnant or breast-feeding patients or women at child-bearing ages without taking acceptable contraceptive measures;
7. Patients received albumin or other blood preparations within 4 days prior to trial drug administration;
8. Patients participated in clinical trials of other drugs within 1 month prior to screening;
9. Patients participated in tolvaptan trials and took tolvaptan previously;
10. Patients are unsuitable to participate in this trial in investigators' opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Body weight changes after 7 days of treatment (quantity of changes) | from day1 to day7

SECONDARY OUTCOMES:
Body weight change after 4 days of treatment (quantity of changes) | from day1 to day4
Waist circumference after 4 and 7 days of treatment (quantity and rate of changes) | from day1 to day7

CONTACTS AND LOCATIONS:
Overall Officials: Minde Zeng, Principal Investigator — RenJi Hospital
Locations (1):
- Renji hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang S, Zhang X, Han T, Xie W, Li Y, Ma H, Liebe R, Weng H, Ding HG. Tolvaptan treatment improves survival of cirrhotic patients with ascites and hyponatremia. BMC Gastroenterol. 2018 Sep 4;18(1):137. doi: 10.1186/s12876-018-0857-0. PMID 30180806